CLINICAL TRIAL: NCT02320071
Title: Abdominal Wall Function and Quality of Life and Before and After Incisional Hernia Repair
Acronym: QualiFunc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, MD, PHD student, Bispebjerg Hospital
Other Study IDs: H-1-2014-118
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with incisional hernia: Patients with one or more incisional hernias, combined horizontal fascial defect 3-8 cm, planned for laparoscopic mesh repair. Patients are examined before and one and three months postoperative in regard to abdominal wall function, pain, discomfort, hernia-related quality of life and physical activity level.
  Interventions: Other: Examination of abdominal wall strength changes over time

INTERVENTIONS:
Other: Examination of abdominal wall strength changes over time

SUMMARY:
The primary objective of the present study is to investigate a possible correlation between abdominal wall function and subjective measures of QoL before and after laparoscopic repair of small- to medium sized incisional hernia.

This prospective study includes 25 patients undergoing laparoscopic incisional hernia repair. Abdominal wall function is examined by determination of maximal truncal flexion and extension with a fixated pelvis using a Goodstrength dynamometer (Metitur Ltd., Jyväskylä, Finland). Subjective scores of QoL (HerQLes), pain (visual analogue scale) and physical activity (International Physical Activity Questionnaire) are assessed. Patients are examined before, one month after and three months after the operation. Furthermore, pulmonary function is examined preoperative and three months postoperative by standard spirometry (forved vital capacity, peak expiratory flow, forced expiratory volume in 1 second) as well as maximum in- and expiratory pressure is measured.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic repair for one or more incisional hernias in the midline (at least 5 cm caudal to the xiphoid process and at least 5 cm cranial to the pubic bone), using a synthetic mesh
* Horizontal fascial defect between 3 and 8 cm
* Age between 25 and 75 years
* American Association of Anesthesiologist score between I and III
* Body mass index < 33 kg/m^2

Exclusion Criteria:

* Severe musculoskeletal, neurologic or cardiopulmonary disease preventing the patient from climbing stairs or shopping for groceries
* Existing stoma
* Postoperative complications requiring intervention

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study includes 25 patients undergoing elective laparoscopic incisional hernia repair. Patients are included from Bispebjerg Hospital and Hvidovre Hospital, two university hospital surgical departments with unrestricted referral of patients.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Abdominal wall strength | Change at three months from baseline examination
  Abdominal wall strength measured by Goodstrength Dynamometer before, one and three months after laparoscopic incisional hernia repair.
Hernia-related quality of life | Change at three months from baseline examination
  Hernia-related quality of life (HerQLes) before, one and three months after laparoscopic incisional hernia repair.

SECONDARY OUTCOMES:
Physical activity level | Change at three months from baseline examination
  International Physical Activity Questionnaire (IPAQ) score before and three months after laparoscopic incisional hernia repair.
Pain | Change at three months from baseline examination
  Pain on visual analogue scale (VAS) before and three months after laparoscopic incisional hernia repair.
Discomfort | Change at three months from baseline examination
  Discomfort on visual analogue scale (VAS) before and three months after laparoscopic incisional hernia repair.
Forced vital capacity | Change at three months from baseline examination
  Forced vital capacity measured by spirometry
Forced expiratorry volume for one second (FEV1) | Change at three months from baseline examination
  Forced expiratorry volume for one second measured by spirometry
Maximal inspiratory pressure | Change at three months from baseline examination
  Maximal inspiratory pressure measured by pressure monitor
Maximal expiratory pressure | Change at three months from baseline examination
  Maximal inspiratory pressure measured by pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, MD, Dr. Msc., Study Chair — Gastrounit, Surgical Section, Hvidovre Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen Northwest, Copenhagen, Denmark